CLINICAL TRIAL: NCT06074341
Title: Mindfulness-Based Relapse Prevention as Video Conferencing Continuing Care to Promote Long Term Recovery From Alcohol Use Disorder
Brief Title: TeleHealth Resources for IndiVidualizEd Goals (THRIVE) in Alcohol Recovery Study
Acronym: THRIVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2212028742; R01AA031159 (NIH)
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder; Alcohol Drinking; Alcohol-Related Disorders
Keywords: mindfulness; recovery; mutual help; harm reduction
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Alcohol-Related Disorders; Harm Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based relapse prevention (Experimental): The MBRP condition will be based on an existing rolling group treatment manual, which consists of eight 60-minute sessions. Each session will begin with a brief mindfulness practice and a discussion of "what is mindfulness?" and the role mindfulness may play in recovery. The themes are repeated every eight sessions, but in every session the participant is bringing a new direct moment experience to the practices in that session. The groups will also consist of people in various stages of recovery and familiarity with the material, which can make for richer discussions of the material led by the group members themselves. Participants who are randomized to receive rolling MBRP treatment will also have access to the Thrive Recovery smart phone app, which includes audio-guided MBRP meditations for participants to practice in daily life.
  Interventions: Behavioral: Mindfulness-based relapse prevention
- Referral to online mutual support groups (Active Comparator): The referral group will consist of a brief 1:1 meeting with a research team member who will provide an orientation to online mutual support and discuss the SMART Recovery, Alcoholics Anonymous (AA), and other virtual meeting options and to discuss how to access mutual support via these platforms. Individuals will also have an opportunity to review the process of attending online groups, and will discuss technology issues that might arise during groups. The session will be 20-30 minutes in length.
  Interventions: Behavioral: Online Mutual Support Groups

INTERVENTIONS:
Behavioral: Mindfulness-based relapse prevention — Mindfulness-based relapse prevention (MBRP) is a group-based treatment to provide individuals with skills intended to foster increased awareness of triggers, destructive habitual patterns, and "automatic" reactions to triggering experiences. Mindfulness practices in MBRP are designed to help individuals pause, observe present experience, and bring awareness to the range of choices available in every moment. Through MBRP individuals learn to respond in ways that serve them, rather than react in ways that are detrimental to their health and happiness.
  Arms: Mindfulness-based relapse prevention
Behavioral: Online Mutual Support Groups — Mutual support groups are free, peer-led organizations that are designed to help individuals with substance use disorders and other addiction-related problems. Mutual support groups often focus on communication and exchange of addiction and recovery experience and skills. Individuals participate in activities that engage, educate, and support patients recovering from substance use disorder from others facing similar challenges. Mutual help organizations that will be offered as referrals include: Alcoholics Anonymous (AA), In The Rooms, and SMART Recovery.
  Arms: Referral to online mutual support groups

SUMMARY:
This project will evaluate the effectiveness and mechanisms of mindfulness-based relapse prevention (MBRP) delivered via video conferencing, as compared to referral to online mutual support groups, in supporting long-term whole-person recovery and improvements in neurobiologically-informed domains of addiction among individuals with alcohol use disorder who are interested in reducing or stopping drinking. The project will also examine the reach, effectiveness, adoption, implementation, and maintenance of MBRP as an accessible and freely available continuing care option that supports long-term recovery from alcohol use disorder in all communities nationwide, including medically underserved and health professional shortage areas.

DETAILED DESCRIPTION:
The goal of this study is to examine the effectiveness of mindfulness-based relapse prevention (MBRP) groups delivered via Zoom in promoting whole-person recovery from alcohol use disorder, and to examine how MBRP affects mechanisms of behavior change based on neurobiologically-informed addiction cycle domains. The investigators will use a hybrid effectiveness-implementation design to prospectively test the effectiveness of MBRP, as well as identify barriers and facilitators of MBRP group participation to inform future implementation of MBRP continuing care. Individuals (n=430) who have recently engaged in a change attempt to stop or reduce their drinking (via treatment or self-change) will be randomized to either MBRP groups via Zoom or referral to online mutual support. Participants will complete measures of psychosocial functioning, alcohol and other drug use, addiction cycle domains, and previously established predictors of recovery every 6 months for 3 years. Using a mixed methods design in the MBRP group, the investigators will examine facilitators and barriers to participation and engagement in MBRP, and assess the reach, effectiveness, adoption, implementation, and maintenance of MBRP via Zoom as continuing care in communities nationwide.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Received AUD treatment or made a self-change attempt to reduce or stop drinking in the past 3 months or is interested in reducing or stopping drinking
* Meet criteria for a current AUD
* Engaged in heavy drinking (more than 14 standard drinks per week or more than 4 drinks on a single day for men and more than 7 drinks per week or more than 3 drinks on a single day for women) in the past 6-months
* Able to understand all study procedures and able to consent in English or Spanish.
* Be willing to use a personal smart phone or tablet that is connected to the internet, or being willing to use a study-provided tablet
* Have access to a valid U.S. mailing address for receiving dried blood spot card or blood collection device.

Exclusion Criteria:

* Current symptoms of psychosis or mania.
* Have a substance use disorder requiring a higher level of care than outpatient treatment (e.g., severe alcohol use disorder requiring inpatient detoxification).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Recovery from AUD | Change from baseline to three year follow-up period
  Recovery is a binary (yes/no) outcome defined by achieving all three of the following: (1) Remission from Diagnostic and Statistical Manual, 5th edition alcohol use disorder (AUD) based on an 11-item AUD symptom checklist (endorsing 0 or 1 item is AUD remission); (2) Cessation of heavy drinking (defined as not engaging in heavy drinking over the past 28 days with heavy drinking defined as 4 or more drinks per occasion for females, and 5 or more drinks per occasion for males, measured by the Timeline Follow-Back); and (3) Improvements in functioning and well-being as measured by higher score on the World Health Organization Quality of Life domain scores (each of 26 items scored from 1 to 5 on a response scale, which are then transformed linearly to a 0-100-scale) and the 36-item Short Form Health Survey Mental Health Component Score (scored on a 0-100 scale). Recovery is achieved if remission, cessation of heavy drinking, and improvements in functioning and well-being are achieved.

SECONDARY OUTCOMES:
Reduction in World Health Organization risk drinking levels | Change from baseline to three year follow-up period
  The Timeline Follow-Back calendar method of assessing standard alcohol drinks consumed each day over the past 28 days will be used to calculate the World Health Organization risk levels based on sex specific grams of alcohol consumed per day in the 28 days prior to the assessment, with levels defined as: low risk (0-20 females/0-40 males), moderate risk (21-40 females, 41-60 males), high risk (41-60 females, 61-100 males), and very high risk (61+ females/100+ males) we will examine those who achieve at least a 1-level and at least a 2-level reduction in risk drinking levels. The reference group for the 1-level reduction is no change or increase in WHO risk drinking level and the reference group for the 2-level reduction is 1-level reduction, no change, or increase in WHO risk drinking level. The Timeline Follow-Back Calendar will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36.
PROMIS Alcohol Negative Consequences | Change from baseline to three year follow-up period
  The Patient-Reported Outcomes Measurement Information System (PROMIS®) includes 7 items scored from never=1 to almost always=5 that assess negative consequences from alcohol use (e.g., I used poor judgment when I drank). The PROMIS Negative Alcohol Consequences measure will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher scores indicate more negative consequences.
PROMIS Preference Score (PROPr) | Change from baseline to three year follow-up period
  PROPr combines scores from 7 PROMIS domains (cognitive function, depression, fatigue, pain interference, physical function, ability to participate in social roles and activities, and sleep disturbance) into a single health utility score. The PROMIS PROPr will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher scores indicate better health.
Penn Alcohol Craving Scale | Change from baseline to three year follow-up period
  Five item measure of overall craving for alcohol. Responses range from 0 to 6 where 0 represents the absence of the specific craving symptom in the item, and 6 represents the maximum intensity or frequency of the craving symptom in the item. The Penn Alcohol Craving Scale will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher scores on the Penn Alcohol Craving Scale reflect more severe alcohol craving.
Alcohol Use Disorder symptoms | Change from baseline to three year follow-up period
  Total number of symptoms endorsed (yes or no) on an 11-item checklist of the symptoms of alcohol use disorder experienced in the past 12-months (baseline) and past 6-months (at 6-month follow-up assessments). The Alcohol Use Disorder Symptom checklist will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher scores indicate more symptoms of alcohol use disorder.
Reduction in percent heavy drinking days | Change from baseline to three year follow-up period
  Percent heavy drinking days will be calculated using the Timeline Follow-Back calendar method of assessing standard alcohol drinks consumed each day over the past 28 days. This measure will be used to identify the total number of occasions of daily heavy drinking (defined as 4 or more drinks for females and 5 or more drinks for males), and the percent heavy drinking days will be calculated as the number of heavy drinking days in the past 28 days divided by the total number of days in that time period (typically 28 days, unless some days are missing). The Timeline Follow-Back Calendar will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher percent heavy drinking days indicate more heavy drinking occasions in a 28-day period.
Reduction in drinks per drinking day | Change from baseline to three year follow-up period
  Drinks per drinking day will be calculated using the Timeline Follow-Back calendar method of assessing standard alcohol drinks consumed each day over the past 28 days. This measure will be used to identify the total number of drinks consumed on each drinking day, and the number of drinks per drinking drinking days will be calculated as the total number of drinks consumed in the past 28 days divided by the total number of days in that time period when drinking occurred (typically 28 days, unless some days are missing). The Timeline Follow-Back Calendar will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher drinks per drinking day indicates greater intensity of drinking in a 28-day period.
Reduction in percent drinking days | Change from baseline to three year follow-up period
  Percent drinking days will be calculated using the Timeline Follow-Back calendar method of assessing standard alcohol drinks consumed each day over the past 28 days. This measure will be used to identify the total number of occasions of drinking, and the percent drinking days will be calculated as the number of drinking days in the past 28 days divided by the total number of days in that time period (typically 28 days, unless some days are missing). The Timeline Follow-Back Calendar will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher percent drinking days indicate greater frequency of drinking in a 28-day period.
World Health Organization Quality of Life (WHOQOL - BREF) Measure | Change from baseline to three year follow-up period
  The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale. The WHOQOL - BREF will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher scores on the WHOQOL-BREF reflect greater quality of life.
Substance Use Moderation Self-Efficacy Scale (SUM-SES) | Change from baseline to three year follow-up period
  The SUM-SES is a 12-item questionnaire that asks participants to indicate on a 0% to 100% scale regarding how confident they are that they would be able to resist drinking beyond their limit in a given situation. The SUM-SES will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher scores on the SUM-SES reflect greater confidence to resist drinking beyond one's limit.
Addiction Cycle - Negative Emotionality Scale | Change from baseline to three year follow-up period
  The negative emotionality domain of the addiction cycle is characterized by temptation to drink in situations when the person is experiencing negative emotions. The Negative Emotionality Scale consists of 4 items scored on a scale from 1=not at all tempted to 5=extremely tempted to drink when experiencing negative emotions. The Addiction Cycle Negative Emotionality scale will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher scores indicate a greater tendency to be tempted to drink in situations characterized by negative emotions.
Addiction Cycle - Incentive Salience Scale | Change from baseline to three year follow-up period
  The incentive salience domain of the addiction cycle is characterized by temptation to drink in situations when the person is experiencing rewarding or social pressure to drink. The Incentive Salience Scale consists of 4 items scored on a scale from 1=not at all tempted to 5=extremely tempted to drink when experiencing rewarding, craving, or social situations. The Addiction Cycle Incentive salience scale will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher scores indicate a greater tendency to be tempted to drink in situations characterized by reward, craving, and social pressure.
Addiction Cycle - Executive Function Scale | Change from baseline to three year follow-up period
  The executive function domain of the addiction cycle is characterized by loss of control over drinking. The Executive Scale consists of 1 binary yes/no item ("After taking one or two drinks, can you usually stop?") and 4 items scored on a scale from 1=indicating more control over drinking to 5=indicating loss of control over drinking. The Addiction Cycle Executive Function scale will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher scores indicate more impaired executive function and greater loss of control over drinking.
Purpose in Life test | Change from baseline to three year follow-up period
  The Purpose in Life test is a 20 item measure of experiencing meaning and purpose in one's life, with each item assessed on a 1 (lack of meaning) to 7 (full of meaning) Likert-type scale. The Purpose in Life test will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher scores indicate more meaning and purpose in life.
PROMIS Meaning and Purpose measure | Change from baseline to three year follow-up period
  The Patient-Reported Outcomes Measurement Information System (PROMIS®) Meaning and Purpose measure includes 8 items scored from not at all=1 to very much=5 that assess one's sense that life has purpose and there are good reasons for living (e.g., My life has meaning). The PROMIS Meaning and Purpose measure will be administered once at baseline, and at follow-up months 6, 12, 18, 24, 30, and 36. Higher scores indicate greater purpose in life

CONTACTS AND LOCATIONS:
Overall Officials: Katie Witkiewitz, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will comply with all NIAAA Data Archives policies established during the project period. This includes compliance with the NIAAA central data platform requirements and timelines developed through the NIAAA Data Share.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the time of publication of the primary manuscript, or within 12 months of last patient assessment.
Access Criteria: Implementation of the plan will follow the NIAAA Data Archive and Data Sharing Policy
URL: https://www.niaaa.nih.gov/research/niaaa-data-archive